CLINICAL TRIAL: NCT02763982
Title: Correlation Between Cardiac Function and Inspiratory Muscles Performance, Chest Wall Volumes and Quality of Life in Individuals With Heart Failure
Brief Title: Cardiac Function and Inspiratory Muscles Performance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Peterson Filipe Pinheiro de Lima, Principal Investigator, Universidade Federal de Pernambuco
Other Study IDs: 39797414.2.0000.520
Record Dates: First submitted 2016-05-02; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure
Keywords: left ventricular ejection fraction; peak oxygen uptake; respiratory muscles; quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- G1: High or normal left ventricular ejection fraction
  Interventions: Other: Physical evaluation
- G2: Moderate left ventricular ejection fraction
  Interventions: Other: Physical evaluation
- G3: Reduced left ventricular ejection fraction
  Interventions: Other: Physical evaluation

INTERVENTIONS:
Other: Physical evaluation

SUMMARY:
The purpose of this study is to determine whether ejection fraction and peak oxygen uptake have correlation on inspiratory muscle strength, chest wall volumes and quality of life in individuals with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Will be included individuals diagnosed with heart failure, both sexes, aged 18-65 years;
* hemodynamically stable (systolic blood pressure ≤ 140 mmHg; diastolic blood pressure ≤ 90 mmHg; heart rate = 90 bpm);
* self-reported sedentary.

Exclusion Criteria:

* Will be excluded individuals with unstable angina were excluded;
* acute myocardial infarction or previous surgery up to three months before the survey;
* musculoskeletal changes, respiratory or chronic metabolic diseases;
* treatment with steroids, hormones or chemotherapy;
* gestation;
* smokers and former smokers assets or liabilities;
* inability to comply with verbal commands appraiser or unsuitability to the evaluation devices.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both female and male participants are being studied, between 18 to 65 years old, diagnosed with heart failure.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Correlation between left ventricular ejection fraction and peak oxygen uptake on inspiratory muscle strength as assessed by echocardiography, ergospirometer and mouth pressure maneuver, respectively | through study completion, an average of 6 months

SECONDARY OUTCOMES:
Correlation between left ventricular ejection fraction and peak oxygen uptake on chest wall volumes as assessed by echocardiography, ergospirometer and opto-electronic plethysmography, respectively | through study completion, an average of 6 months
Correlation between left ventricular ejection fraction and peak oxygen uptake on quality of life as assessed by echocardiography, ergospirometer and Minnesota Living with Heart Failure Questionnaire, respectively | through study completion, an average of 6 months

REFERENCES:
- [Result] Yamada K, Kinugasa Y, Sota T, Miyagi M, Sugihara S, Kato M, Yamamoto K. Inspiratory Muscle Weakness is Associated With Exercise Intolerance in Patients With Heart Failure With Preserved Ejection Fraction: A Preliminary Study. J Card Fail. 2016 Jan;22(1):38-47. doi: 10.1016/j.cardfail.2015.10.010. Epub 2015 Oct 23. PMID 26505812
- [Result] Verissimo P, Casalaspo TJ, Goncalves LH, Yang AS, Eid RC, Timenetsky KT. High prevalence of respiratory muscle weakness in hospitalized acute heart failure elderly patients. PLoS One. 2015 Feb 11;10(2):e0118218. doi: 10.1371/journal.pone.0118218. eCollection 2015. PMID 25671566
- [Result] Adamopoulos S, Schmid JP, Dendale P, Poerschke D, Hansen D, Dritsas A, Kouloubinis A, Alders T, Gkouziouta A, Reyckers I, Vartela V, Plessas N, Doulaptsis C, Saner H, Laoutaris ID. Combined aerobic/inspiratory muscle training vs. aerobic training in patients with chronic heart failure: The Vent-HeFT trial: a European prospective multicentre randomized trial. Eur J Heart Fail. 2014 May;16(5):574-82. doi: 10.1002/ejhf.70. Epub 2014 Mar 14. PMID 24634346
- [Result] Stamm O, Latscha U, Janecek P, Campana A. Development of a special electrode for continuous subcutaneous pH measurement in the infant scalp. Am J Obstet Gynecol. 1976 Jan 15;124(2):193-5. doi: 10.1016/s0002-9378(16)33297-5. PMID 2012